CLINICAL TRIAL: NCT03425019
Title: Self Transcranial Direct Current Stimulation for Pain in Older Adults With Knee Osteoarthritis (Self tDCS and Knee Pain)
Brief Title: Self Transcranial Direct Current Stimulation for Pain in Older Adults With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Hyochol Ahn, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SN-17-1072
Record Dates: First submitted 2018-01-30; First posted 2018-02-07 (Actual); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Knee Osteoarthritis; Chronic Pain
Keywords: Knee Osteoarthritis; Chronic Pain; Osteoarthritis; Transcranial Direct Current Stimulation; tDCS
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Transcranial Direct Current Stimulation (Experimental): Transcranial Direct Current Stimulation (tDCS) involves the application of weak direct electric current to the head in a noninvasive and painless manner. tDCS with a constant current intensity of 2 milliamps (mA) will be applied for 20 minutes per session daily for 2 weeks (Monday to Friday) via the Soterix 1x1 tDCS mini-CT Stimulator device. Participants will self-administer tDCS at their home or a private room for two weeks (Mondays-Fridays) under real-time supervision by the research staff.
  Interventions: Device: Soterix 1x1 tDCS mini-CT Stimulator device

INTERVENTIONS:
Device: Soterix 1x1 tDCS mini-CT Stimulator device — Transcranial Direct Current Stimulation (tDCS) involves the application of weak direct electric current to the head in a noninvasive and painless manner. tDCS with a constant current intensity of 2 mA will be applied for 20 minutes per session daily for 2 weeks (Monday to Friday) via the Soterix 1x1 tDCS mini-CT Stimulator device. Participants will self-administer tDCS at their home or a private room for two weeks (Mondays-Fridays) under real-time supervision by the research staff.

SUMMARY:
The purpose of this study is to determine the feasibility and preliminary efficacy of two weeks of self Transcranial Direct Current Stimulation (tDCS) for pain in older patients with knee osteoarthritis (OA).

ELIGIBILITY:
Inclusion Criteria:

* have self-reported unilateral or bilateral knee OA pain, according to American College of Rheumatology criteria
* have had knee OA pain in the past 3 months with an average of at least 3 on a 10 cm Visual Analog Scale (VAS) for pain
* can speak and read English
* have a device with internet access that can be used for secure video conferencing for real-time remote supervision
* have access to a distraction-free, well lit, clean environment with a safe area to store the device and device kit
* have no plan to change medication regimens for pain throughout the trial
* are able to travel to the coordinating center
* are willing and able to provide written informed consent prior to enrollment.

Exclusion Criteria:

* previous prosthetic knee replacement or non-arthroscopic surgery to the affected knee
* history of brain surgery, tumor, seizure, stroke, or intracranial metal implantation
* systemic rheumatic disorders, including rheumatoid arthritis, systemic lupus erythematosus, and fibromyalgia
* uncontrolled hypertension (i.e., systolic blood pressure/ diastolic blood pressure ≥ 150/95 mm Hg)
* heart failure
* history of acute myocardial infarction
* peripheral neuropathy
* alcohol/substance abuse
* cognitive impairment (i.e., Mini-Mental Status Exam score ≤ 23)
* pregnancy or lactation
* hospitalization within the preceding year for psychiatric illness

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyochol Ahn, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahn H, Sorkpor S, Miao H, Zhong C, Jorge R, Park L, Abdi S, Cho RY. Home-based self-administered transcranial direct current stimulation in older adults with knee osteoarthritis pain: An open-label study. J Clin Neurosci. 2019 Aug;66:61-65. doi: 10.1016/j.jocn.2019.05.023. Epub 2019 May 29. PMID 31153751

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant withdrew before the intervention started.
Groups:
- Transcranial Direct Current Stimulation: Transcranial Direct Current Stimulation (tDCS) involves the application of weak direct electric current to the head in a noninvasive and painless manner. tDCS with a constant current intensity of 2 mA will be applied for 20 minutes per session daily for 2 weeks (Monday to Friday) via the Soterix 1x1 tDCS mini-CT Stimulator device. Participants will self-administer tDCS at their home or a private room for two weeks (Mondays-Fridays) under real-time supervision by the research staff.
Period: Overall Study
Arm/Group | Transcranial Direct Current Stimulation
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (7.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 6
  Asian | 6
  Hispanic | 1
  White | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Education [Count of Participants; unit: Participants]
  High School | 3
  2-year college | 5
  4-year college | 9
  Master's degree | 2
  Doctoral degree | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.33 (8.01)
Osteoarthritis duration [Mean (Standard Deviation); unit: months] | 29.60 (26.17)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Pain Intensity as Assessed by a Visual Analogue Scale (VAS)
Description: Scores on the visual analogue scale (VAS) range from 0 (no pain) to 100 (worst pain imaginable).
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 55.23 (25.45)

2. Primary Outcome: Clinical Pain Intensity as Assessed by a Visual Analogue Scale (VAS)
Description: Scores on the visual analogue scale (VAS) range from 0 (no pain) to 100 (worst pain imaginable).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 24.85 (22.70)

3. Secondary Outcome: Clinical Pain Intensity as Assessed by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) - Pain Subscale
Description: The WOMAC is a self-administered questionnaire consisting of 3 subscales related to pain (pain subscale total score range, 0-20), stiffness (stiffness subscale total score range, 0-8), and impairments of physical function (functional impairment subscale range, 0-68), with higher scores indicating worse pain, stiffness, and impairments of physical function, respectively.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
score on a scale | 7.95 (4.39)

4. Secondary Outcome: Clinical Pain Intensity as Assessed by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) - Pain Subscale
Description: as for outcome 3
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 5.75 (4.25)

5. Secondary Outcome: Clinical Pain Intensity as Assessed by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) - Stiffness Subscale
Description: as for outcome 3
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 4.00 (1.86)

6. Secondary Outcome: Clinical Pain Intensity as Assessed by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) - Stiffness Subscale
Description: as for outcome 3
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 2.90 (1.74)

7. Secondary Outcome: Clinical Pain Intensity as Assessed by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) - Functional Impairment Subscale
Description: as for outcome 3
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 29.10 (17.53)

8. Secondary Outcome: Clinical Pain Intensity as Assessed by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) - Functional Impairment Subscale
Description: as for outcome 3
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 20.85 (15.22)

9. Secondary Outcome: Clinical Pain Intensity as Assessed by Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) - Continuous Pain Summary Scale
Description: The SF-MPQ-2 measures the quality as well as the intensity of pain. Participants complete the SF-MPQ-2 by rating the extent to which they experienced each of 22 pain descriptors in the past week using an 11-point numeric rating scale (0 = "none" to 10 = "worst possible"). The continuous pain subscale assesses throbbing pain, cramping pain, gnawing pain, aching pain, heavy pain, and tender, and total score on the continuous pain subscale ranges from 0-60, with a higher score indicating worse pain.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 22.75 (15.26)

10. Secondary Outcome: Clinical Pain Intensity as Assessed by Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) - Continuous Pain Subscale
Description: as for outcome 9
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 14.05 (13.84)

11. Secondary Outcome: Clinical Pain Intensity as Assessed by Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) - Intermittent Pain Subscale
Description: The SF-MPQ-2 measures the quality as well as the intensity of pain. Participants complete the SF-MPQ-2 by rating the extent to which they experienced each of 22 pain descriptors in the past week using an 11-point numeric rating scale (0 = "none" to 10 = "worst possible"). The intermittent pain subscale assesses shooting pain, stabbing pain, sharp pain, splitting pain, electric-shock pain, and piercing, and total score on the intermittent pain subscale ranges from 0-60, with a higher score indicating worse pain.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 17.80 (16.18)

12. Secondary Outcome: Clinical Pain Intensity as Assessed by Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) - Intermittent Pain Subscale
Description: as for outcome 11
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 12.90 (15.80)

13. Secondary Outcome: Clinical Pain Intensity as Assessed by Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) - Neuropathic Pain Subscale
Description: The SF-MPQ-2 measures the quality as well as the intensity of pain. Participants complete the SF-MPQ-2 by rating the extent to which they experienced each of 22 pain descriptors in the past week using an 11-point numeric rating scale (0 = "none" to 10 = "worst possible"). The neuropathic pain subscale assesses hot-burning pain, cold-freezing pain, pain caused by light touch, itching, tingling or 'pins and needles', and numbness, and total score on the neuropathic pain subscale ranges from 0-60, with a higher score indicating worse pain.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 11.1 (13.71)

14. Secondary Outcome: Clinical Pain Intensity as Assessed by Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) - Neuropathic Pain Subscale
Description: as for outcome 13
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 8.2 (14.23)

15. Secondary Outcome: Clinical Pain Intensity as Assessed by Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) - Affective Description Subscale
Description: The SF-MPQ-2 measures the quality as well as the intensity of pain. Participants complete the SF-MPQ-2 by rating the extent to which they experienced each of 22 pain descriptors in the past week using an 11-point numeric rating scale (0 = "none" to 10 = "worst possible"). The affective description subscale assesses tiring-exhausting, sickening, fearful, and punishing-cruel, and total score on the affective description subscale ranges from 0-40, with a higher score indicating worse pain.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 11.7 (11.65)

16. Secondary Outcome: Clinical Pain Intensity as Assessed by Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) - Affective Description Subscale
Description: as for outcome 15
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 5.75 (10.40)

17. Secondary Outcome: Experimental Pain Sensitivity as Assessed by a Multimodal Quantitative Sensory Testing (QST) Battery - Heat Pain Threshold (HPTH)
Description: In order to measure experimental pain sensitivity, a multimodal Quantitative Sensory Testing (QST) battery will be completed: heat pain threshold (HPTH); heat pain tolerance (HPTO), pressure pain threshold (PPT), punctate mechanical pain (PMP), and Conditioned Pain Modulation (CPM).
  To assess HPTH, heat stimuli were delivered to the participant's arm or knee using a computer-controlled TSAII NeuroSensory Analyzer. From a baseline of 32 degrees Celsius, the temperature increased by 0.5 degrees Celsius per second until the participants responded by pressing a button to stop heat stimuli. Participants were instructed to press the button when the sensation ''first becomes painful" to assess the heat pain threshold (HPTH). The temperature at which participants pressed the button to indicate the sensation ''first becomes painful" is reported.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
degrees Celsius
  arm | 37.9 (3.3)
  knee | 39.1 (3.5)

18. Secondary Outcome: Experimental Pain Sensitivity as Assessed by a Multimodal Quantitative Sensory Testing (QST) Battery - Heat Pain Threshold (HPTH)
Description: as for outcome 17
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
degrees Celsius
  arm | 37.3 (2.0)
  knee | 40.1 (3.4)

19. Secondary Outcome: Experimental Pain Sensitivity as Assessed by a Multimodal Quantitative Sensory Testing (QST) Battery - Heat Pain Tolerance (HPTO)
Description: In order to measure experimental pain sensitivity, a multimodal Quantitative Sensory Testing (QST) battery will be completed: heat pain threshold (HPTH); heat pain tolerance (HPTO), pressure pain threshold (PPT), punctate mechanical pain (PMP), and Conditioned Pain Modulation (CPM).
  To assess HPTO, heat stimuli were delivered to the participant's arm or knee using a computer-controlled TSAII NeuroSensory Analyzer. From a baseline of 32 degrees Celsius, the temperature increased by 0.5 degrees Celsius per second until the participants responded by pressing a button to stop heat stimuli. Participants were instructed to press the button when they ''no longer feel able to tolerate the pain." The temperature at which participants pressed the button to indicate they could ''no longer feel able to tolerate the pain" is reported.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
degrees Celsius
  arm | 43.2 (3.1)
  knee | 43.1 (3.3)

20. Secondary Outcome: Experimental Pain Sensitivity as Assessed by a Multimodal Quantitative Sensory Testing (QST) Battery - Heat Pain Tolerance (HPTO)
Description: as for outcome 19
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
degrees Celsius
  arm | 43.2 (3.2)
  knee | 44.6 (3.1)

21. Secondary Outcome: Experimental Pain Sensitivity as Assessed by a Multimodal Quantitative Sensory Testing (QST) Battery - Pressure Pain Threshold (PPT)
Description: In order to measure experimental pain sensitivity, a multimodal Quantitative Sensory Testing (QST) battery will be completed: heat pain threshold (HPTH); heat pain tolerance (HPTO), pressure pain threshold (PPT), punctate mechanical pain (PMP), and Conditioned Pain Modulation (CPM).
  To assess PPT, a handheld digital pressure algometer (Wagner, Greenwich, CT) was applied at a constant rate of 0.3 kilograms force per centimeter squared (kgf/cm^2) per second to the participant's medial knee, lateral knee, or trapezius. Participants were asked to notify the experimenter when the pressure sensation ''first becomes painful." The pressure at which participants pressed the button to indicate that the pressure sensation ''first becomes painful" is reported.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: kilograms force (kgf)
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
kilograms force (kgf)
  medial knee | 3.2 (1.4)
  lateral knee | 3.5 (1.5)
  trapezius | 2.9 (1.6)

22. Secondary Outcome: Experimental Pain Sensitivity as Assessed by a Multimodal Quantitative Sensory Testing (QST) Battery - Pressure Pain Threshold (PPT)
Description: as for outcome 21
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: kilograms force (kgf)
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
kilograms force (kgf)
  medial knee | 3.7 (1.2)
  lateral knee | 4.4 (1.3)
  trapezius | 3.9 (1.3)

23. Secondary Outcome: Experimental Pain Sensitivity as Assessed by a Multimodal Quantitative Sensory Testing (QST) Battery - Punctate Mechanical Pain (PMP)
Description: In order to measure experimental pain sensitivity, a multimodal Quantitative Sensory Testing (QST) battery will be completed: heat pain threshold (HPTH); heat pain tolerance (HPTO), pressure pain threshold (PPT), punctate mechanical pain (PMP), and Conditioned Pain Modulation (CPM).
  To assess PMP, punctate mechanical pain is delivered to the patella or hand by a calibrated nylon monofilament for 10 contacts of the monofilament at one contact per second. Participants rate the pain intensity on a scale from 0 (no pain) to 100 (maximum imaginable pain).
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
score on a scale
  patella | 84.7 (23.4)
  hand | 66.0 (27.0)

24. Secondary Outcome: Experimental Pain Sensitivity as Assessed by a Multimodal Quantitative Sensory Testing (QST) Battery - Punctate Mechanical Pain (PMP)
Description: as for outcome 23
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
score on a scale
  patella | 67.4 (26.9)
  hand | 54.6 (23.9)

25. Secondary Outcome: Experimental Pain Sensitivity as Assessed by a Multimodal Quantitative Sensory Testing (QST) Battery - Conditioned Pain Modulation (CPM)
Description: In order to measure experimental pain sensitivity, a multimodal Quantitative Sensory Testing (QST) battery will be completed: heat pain threshold (HPTH); heat pain tolerance (HPTO), pressure pain threshold (PPT), punctate mechanical pain (PMP), and Conditioned Pain Modulation (CPM).
  CPM is reported as the change in PPT before and immediately following immersion of the contralateral hand up to the wrist in a cold water bath (12 degrees Celsius) for up to one minute. To assess PPT, a handheld digital pressure algometer (Wagner, Greenwich, CT) was applied at a constant rate of 0.3 kilograms force per centimeter squared (kgf/cm^2) per second to the participant's trapezius. Participants were asked to notify the experimenter when the pressure sensation ''first becomes painful." The pressure at which participants pressed the button to indicate that the pressure sensation ''first becomes painful" is reported.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: kilograms force (kgf)
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
kilograms force (kgf) | 0.9 (0.7)

26. Secondary Outcome: Experimental Pain Sensitivity as Assessed by a Multimodal Quantitative Sensory Testing (QST) Battery - Conditioned Pain Modulation (CPM)
Description: as for outcome 25
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: kilograms force (kgf)
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
kilograms force (kgf) | 1.3 (0.6)

27. Secondary Outcome: Number of Participants Who Were Assessed by Functional Near-infrared Spectroscopy (fNIRS)
Description: Pain-related cortical response will be measured using a continuous-wave, multichannel fNIRS imaging system (LIGHTNIRS, Shimadzu, Kyoto, Japan) with three semiconductor lasers at 780, 805, and 830 nm. Optical recordings will be collected during thermal pain stimulation.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
Participants | 20

28. Secondary Outcome: Feasibility as Assessed by a Survey of Participants' tDCS Experience - Ease of Using Device
Description: Data will be collected on participants' tDCS experience at the conclusion of tDCS treatment on a scale of 0 (strongly disagree) to 10 (strongly agree): Q1) "Overall the device was easy to use"
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
score on a scale | 9.75 (0.44)

29. Secondary Outcome: Feasibility as Assessed by a Survey of Participants' tDCS Experience - Ease of Preparation of Device
Description: Data will be collected on participants' tDCS experience at the conclusion of tDCS treatment on a scale of 0 (strongly disagree) to 10 (strongly agree): Q2) "It was easy to prepare the device and accessories"
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
score on a scale | 9.75 (0.44)

30. Secondary Outcome: Feasibility as Assessed by a Survey of Participants' tDCS Experience - Effectiveness of Treatment Over Time
Description: Data will be collected on participants' tDCS experience at the conclusion of tDCS treatment on a scale of 0 (strongly disagree) to 10 (strongly agree): Q3) "The effectiveness of the treatment increased over the course of treatment."
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
score on a scale | 6.75 (3.17)

31. Secondary Outcome: Tolerability as Assessed by Number of Participants With Side Effects
Description: The participants will be asked in an open-ended manner whether they have experienced any side effects, and they will then be asked specifically about tingling, itching sensation, burning sensation, pain at the stimulation site, fatigue, nervousness, headache, difficulty concentrating, mood change, and changes in vision or visual perception.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
Participants | 0

32. Secondary Outcome: Anxiety as Assessed by the PROMIS Anxiety-short Form
Description: The 7-item PROMIS anxiety-short form assesses the pure domain of anxiety in individuals age 18 and older, and each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 7 to 35 with higher scores indicating greater severity of anxiety.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
score on a scale | 13.6 (6.73)

33. Secondary Outcome: Anxiety as Assessed by the PROMIS Anxiety-short Form
Description: as for outcome 32
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
score on a scale | 12.05 (6.86)

34. Secondary Outcome: Depression as Assessed by the PROMIS Depression-short Form
Description: The 8-item PROMIS depression-short form assesses the pure domain of depression in individuals age 18 and older, and each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of depression.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 12.3 (7.69)

35. Secondary Outcome: Depression as Assessed by the PROMIS Depression-short Form
Description: as for outcome 34
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 11.85 (6.98)

36. Secondary Outcome: Sleep Disturbance as Assessed by the PROMIS Sleep Disturbance-short Form
Description: The 8-item PROMIS sleep disturbance-short form assesses the pure domain of sleep disturbance in individuals age 18 and older, and each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 24.3 (7.87)

37. Secondary Outcome: Sleep Disturbance as Assessed by the PROMIS Sleep Disturbance-short Form
Description: as for outcome 36
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 20
units on a scale | 19.85 (8.10)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Transcranial Direct Current Stimulation
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT03425019/Prot_SAP_000.pdf